CLINICAL TRIAL: NCT06515925
Title: Phase II: GEMINI: Virtual Integrative Medical Group Visits for Managing Chronic Pain
Brief Title: Our Whole Lives Gemini: Virtual Integrative Medical Group Visits for Managing Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); BrightOutcome (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CHA-IRB-23-24-260; 1R44AT012302-01A1 (NIH)
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Our Whole Lives (OWL) (Experimental): Our Whole Lives (OWL) is a 9-week online curriculum on the GEMINI platform. OWL is a nine-session, web-accessible, self-paced mindfulness curriculum that has interactive components of self-monitoring and social support (online community).
  Interventions: Behavioral: Our Whole Lives (OWL)
- Low Dose Mindfulness Training (Active Comparator): The GEMINI platform will facilitate the delivery of a low-dose mindfulness version of Our Whole Lives program. Participants will interface with the GEMINI platform's static content.
  Interventions: Behavioral: Low Dose Mindfulness Training

INTERVENTIONS:
Behavioral: Our Whole Lives (OWL) — OWL is a nine-session, web-accessible, self-paced mindfulness curriculum that has interactive components of self-monitoring and social support (online community). Our Whole Lives (OWL) online curriculum of self-management topics such as mindfulness, mind-body practices, education about chronic pain therapies, stress reduction, sleep, and nutrition.
  Once a week for 9 weeks participants will attend a 1.5 -2-hour online group session via Zoom or Google Meets, accessing it through GEMINI platform.
  Arms: Our Whole Lives (OWL)
Behavioral: Low Dose Mindfulness Training — The GEMINI platform will facilitate the delivery of a low-dose version of Our Whole Lives program. OWL in this arm is a nine-session, web-accessible, self-paced curriculum, self-monitoring. Participants will interface with the GEMINI platform's static content.
  Other Names: Low dose comparator
  Arms: Low Dose Mindfulness Training

SUMMARY:
The goal of this research study is to test the efficacy of a non-prescription medicine, web-based platform solution for patients with chronic pain, to improve pain self-management and related outcomes. The main question investigators aim to answer is; would the use of this web-based intervention plus an online group visit compared to control result in better pain-related outcomes and improved pain impact?

DETAILED DESCRIPTION:
This study has 6 mandatory components and 1 optional component:

* Recruitment Screening Call
* Informed Consent Session
* Baseline Survey Session
* Intervention: Engagement with the Our Whole Lives (OWL) an e-health platform: For 9 weeks, participants will all have access to a mindfulness program within OWL, optimized for people with chronic pain.
* Live-Online Mindfulness Group weekly
* Control: Low dose engagement with OWL with no group engagement.
* Follow-Up Survey Sessions at Week 10, Week 16, and Week 24.
* Online Focus Group/Individual Interview. Participants will be asked to participate in an OPTIONAL individual interview, or a one-hour focus group with other participants in the study who used the OWL website as well.

Researchers will compare two groups that will be using the web-based platform. Each group will have different engagement content from the web-based platform and investigators will see if it affects overall chronic pain and pain management.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults
* Over the age of 18
* Experiencing chronic musculoskeletal pain. (Pain may have more than one source; Pain must be non-malignant; Participant must have an average pain intensity of ≥ 4 (1 out of 10) in the past 7 days; Participant must meet the chronic criteria of a pain problem that has persisted at least 3 months, and has resulted in pain on at least half the days in the past 6 months)

Exclusion Criteria:

* Inability to understand English at a level necessary for informed consent and understanding participation instructions, and participating in the group;
* Serious underlying systemic or co-morbid conditions or life event that precludes physical or cognitive ability to participate in the study.
* Severe depression
* Current mania or psychosis;
* Active heroin or cocaine use in the past 3 months
* Heavy alcohol use
* Known or planned pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Reduced pain impact (based on PROMIS 29) | up to 24 weeks
  The primary trial aim is to reduce pain impact.

SECONDARY OUTCOMES:
The Patient-Reported Outcomes Measurement Information System (PROMIS 29) | up to 24 weeks
  Depression and Anxiety in the past 7 days. Fatigue in the past 7 days. Sleep disturbance in the past 7 days. Ability to Participate in Social roles, and activities. Each item within is measured on a 5-point scale, 1 (minimum) to 5(maximum). Higher T-scores in some domains indicate better health; in others, they indicate worse symptoms.
Pain Self- Efficacy Scale (PSEQ) | up to 24 weeks
  Self-efficacy beliefs for pain management. 10 items measured on a 6-point scale, 0 (minimum) to 6(maximum). Higher scores indicate greater pain self-efficacy.
Timeline Follow-Back (TLFB) | up to 24 weeks
  Use of pain meds in the previous 7 days, including opioid use.

CONTACTS AND LOCATIONS:
Overall Officials: Zev Schuman-Olivier, MD, Study Director — Cambridge Health Alliance; Paula Gardiner, MD, MPH, Principal Investigator — Cambridge Health Alliance; Niina Haas, PHD, Principal Investigator — BrightOutcome
Locations (1):
- Cambridge Health Alliance Center for Mindfulness and Compassion, Malden, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on research standards for chronic low back pain. J Pain. 2014 Jun;15(6):569-85. doi: 10.1016/j.jpain.2014.03.005. Epub 2014 Apr 29. PMID 24787228
- [Background] Deyo RA, Katrina Ramsey, Buckley DI, Michaels L, Kobus A, Eckstrom E, Forro V, Morris C. Performance of a Patient Reported Outcomes Measurement Information System (PROMIS) Short Form in Older Adults with Chronic Musculoskeletal Pain. Pain Med. 2016 Feb;17(2):314-24. doi: 10.1093/pm/pnv046. PMID 26814279
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Sobell LC, Sobell MB. Timeline follow-back. Measuring alcohol consumption. Springer;1992:41-72.
- [Background] Fals-Stewart W, O'Farrell TJ, Freitas TT, McFarlin SK, Rutigliano P. The timeline followback reports of psychoactive substance use by drug-abusing patients: psychometric properties. J Consult Clin Psychol. 2000 Feb;68(1):134-44. doi: 10.1037//0022-006x.68.1.134. PMID 10710848

DOCUMENTS (1):
  • Informed Consent Form (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT06515925/ICF_000.pdf